CLINICAL TRIAL: NCT02474589
Title: An Expanded Double-Blind, Placebo Controlled, Multicenter Trial to Assess the Safety, Tolerability, and Pharmacokinetics of the Anti Orthopoxvirus Compound Tecovirimat When Administered Orally for 14 Days in Subjects
Brief Title: A Trial to Assess the Safety, Tolerability, and Pharmacokinetics of the Anti-Orthopoxvirus Compound Tecovirimat
Acronym: SIGA246-008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIGA-246-008
Record Dates: First submitted 2015-06-01; First posted 2015-06-18 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Smallpox
Keywords: Treatment; orthopoxvirus; smallpox
MeSH Terms: conditions — Smallpox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): 600 mg tecovirimat capsules BID to assess safety and tolerability and pharmacokinetics of the anit-orthopoxvirus compound Tecovirimat when administered orally in healthy subjects
  Interventions: Drug: tecovirimat
- Placebo (Placebo Comparator): matching placebo capsules BID to assess safety and tolerability and pharmacokinetics of the anit-orthopoxvirus compound Tecovirimat when administered orally in healthy subjects
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tecovirimat — Study is based on Animal Regulatory Rule
  Other Names: ST-246
  Arms: Active
Other: Placebo — Does not apply
  Arms: Placebo

SUMMARY:
Multicenter, double-blind, placebo controlled, Phase 3 study to determine the safety and tolerability of oral tecovirimat, an anti orthopoxvirus compound, in subjects.

DETAILED DESCRIPTION:
Pharmacokinetics and safety and tolerability data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old, inclusive
* Available for clinical follow-up for the duration of the study
* Able and willing to give informed consent
* In good general health without clinically significant medical history; not have been hospitalized for a chronic medical condition for the last 2 years
* Able to comply with dietary requirements throughout the study drug dosing period
* Adequate venous access for those individuals participating in PK testing
* PE and laboratory results without clinically significant findings within the 14 days before receipt of study drug
* Agree not to drink alcohol from the beginning of the Screening Period through the completion of the Day 28 Follow up Visit
* Agree not to use any nicotine products, including electronic vapor cigarettes, nicotine patches or nicotine gum for at least 30 days before the Day 1 Visit and through completion of the Day 15 Dosing complete Visit
* Agree not to consume caffeine during all study visits, including overnight stays if participating in PK subset
* Agree not to receive any immunizations/vaccinations
* Agree not to take herbal products
* Able and willing to refrain from taking any prescriptions and nonprescription medications with exceptions
* For women of childbearing potential, negative serum and urine pregnancy testing
* If male, agree not to donate sperm
* Meet 1 of the following criteria: The subject or their partner has undergone surgical sterilization; the subject is postmenopausal; the subject agrees to be abstinent; the subject agrees to consistently use a method of approved birth control.

Exclusion Criteria:

* Pregnant or breast-feeding or planning pregnancy
* Have a history of any clinically significant conditions
* Have any limitation of activity related to cardiac disease
* Have a bleeding disorder diagnosed by a doctor, or a history of significant bruising or bleeding with intramuscular injections or blood draws
* Currently using certain medications
* Have a malignancy that is active or a treated malignancy for which there is no reasonable assurance of sustained cure, or malignancy that is likely to recur during the study
* Have a history of seizure
* Have a clinically significant blood dyscrasia
* Have a history of drug allergy that contraindicates participation in the trial
* Have a medical, psychiatric, or social condition or any occupational reason, or other responsibility that in the judgment of the investigator would render the subject unable to comply with the protocol
* Have an inability to swallow medication
* Have a clinically significant abnormal ECG
* Have participated in a clinical trials within 30 days of study entry or planning to participate in any experimental treatment study during the study period
* Have a history or current drug or alcohol abuse
* Have received immunizations/vaccines
* Have a current clinically significant acute bacterial, fungal, or mycobacterial infection requiring administration of systemic antibiotics
* Have known chronic bacterial, mycobacterial, fungal, parasitic, or protozoal infection with the exception of clinically significant dermal infections
* Have known hepatitis B or C infection, or positive test result
* Have known HIV infection or AIDS or a positive test for HIV
* Have a current clinically significant viral infection
* Have known clinically significant chronic viral infection
* have received treatment with greater than 20 mg prednisone or equivalent dose or any immunosuppressant or immunomodulary medication
* Have abnormal laboratory testing during screening
* Have a greater than or equal than 20% risk of suffering a major cardiovascular event
* Have been previously enrolled in this or any clinical trial involving tecovirimat

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hruby, Ph.D., Study Director — SIGA Technologies, Inc.
Locations (11):
- United States (11):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Paradigm Research, Redding, California
  - Paradigm Research, San Diego, California
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research LLC, St Louis, Missouri
  - Meridien Clinical Research, Omaha, Nebraska
  - Medical Research South, Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grosenbach DW, Honeychurch K, Rose EA, Chinsangaram J, Frimm A, Maiti B, Lovejoy C, Meara I, Long P, Hruby DE. Oral Tecovirimat for the Treatment of Smallpox. N Engl J Med. 2018 Jul 5;379(1):44-53. doi: 10.1056/NEJMoa1705688. PMID 29972742

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 359 | 90
Completed | 334 | 85
Not Completed | 25 | 5
Not completed — Adverse Event | 6 | 2
Not completed — Lost to Follow-up | 6 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Inability to complete study procedures | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 359 | 90 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (15.67) | 41.9 (15.85) | 40.7 (15.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 54 | 265
  Male | 148 | 36 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 5 | 48
  Not Hispanic or Latino | 315 | 85 | 400
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 101 | 26 | 127
  White | 249 | 62 | 311
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 359 | 90 | 449

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Number of Participants With Adverse Events
Description: To determine the safety and tolerability of oral tecovirimat
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 359 | 90
Participants | 134 | 30

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 1 Randomization Visit after study drug dosing through the Day 28 Follow-up Visit. Subjects with unresolved AE/SAE at the Day 28 Follow-up Visit were required to complete a Day 45 AE/SAE only Follow up Visit. All AEs/SAEs were to be followed until the subject was no longer participating in the study, or the AE/SAE was stable or until resolution.
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 1/359 | 0/90
Other Adverse Events (participants affected / at risk) | 134/359 | 30/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=359) | Placebo (N=90)
Pulmonary embolus (pulmonary embolism) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=359) | Placebo (N=90)
Headache (Nervous system disorders) | 61 (104) | 13 (19)
Nausea (Gastrointestinal disorders) | 20 (29) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 3 (4)
Dizziness (Nervous system disorders) | 9 (9) | 3 (3)
Fatigue (General disorders) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 9 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Disturbance in Attention (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (7) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal DIscomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chapped Lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palpable Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis Generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Ligament Sprain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Libido Increased (Psychiatric disorders) | 0 (0) | 1 (1)
Nighmare (Psychiatric disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pumonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sputum Retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vasomotor Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood Pressure Systolic Increased (Investigations) | 2 (2) | 0 (0)
Electroencephalogram Abnormal (Investigations) | 1 (1) | 0 (0)
Haematocrit Decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Menstruation Irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peripheral Coldness (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less